CLINICAL TRIAL: NCT02170129
Title: Sinus Lift Grafting With Anorganic Bovine Bone vs 50% Autologous + 50% Bovine Bone. One Year Results From a Randomized Controlled Trial.
Brief Title: SINUS LIFT 100% Anorganic Bovine Bone vs. 50% Anorganic Bovine Bone + 50% Autologous Bone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Sassari (Other)
Responsible Party: Principal Investigator, Silvio Mario Meloni, DDS, Phd, MS, Università degli Studi di Sassari
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SINUS LIFT
Record Dates: First submitted 2014-06-10; First posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Maxillary Sinus; Dental Implants

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 100% AAB (Active Comparator): Surgical procedures were performed according to a lateral approach technique at the edentulous region distal to the position of the first premolar. A mucoperiosteal buccal flap was elevated, exposing the lateral bony wall of the sinus antrum. A round diamond bur, 2 mm in diameter, was used to outline the demarcation of the lateral window, which was removed, thus completely exposing the underlying Schneiderian membrane. The membrane was separated from the housing bone, and a tension-free reflection exposing the sinus walls was achieved by gently pushing it away using a large flat curette (Kramer-Nevins, Hu-Friedy, Chicago, IL). The established voids were then filled with 100% AAB (Bio-Oss) followed by sealing the open lateral window by the placement of a collagen membrane (Bio Gide) and primary soft tissue closure using Vicryl 4.0 sutures (Vicryl, Ethicon J&J International, Sint-Stevens-Woluwe, Belgium).
  Interventions: Device: 100% AAB
- 50% AAB plus 50% autologous bone (Active Comparator): Surgical procedures were performed according to a lateral approach technique at the edentulous region distal to the position of the first premolar. A mucoperiosteal buccal flap was elevated, exposing the lateral bony wall of the sinus antrum. A round diamond bur, 2 mm in diameter, was used to outline the demarcation of the lateral window, which was removed, thus completely exposing the underlying Schneiderian membrane. The membrane was separated from the housing bone, and a tension-free reflection exposing the sinus walls was achieved by gently pushing it away using a large flat curette (Kramer-Nevins, Hu-Friedy, Chicago, IL). The established voids were then filled with 50% AAB (Bio-Oss) plus 50% autologous bone harvested locally with a bone scraper followed by sealing the open lateral window by the placement of a collagen membrane (Bio Gide) and primary soft tissue closure using Vicryl 4.0 sutures (Vicryl, Ethicon J&J International, Sint-Stevens-Woluwe, Belgium).
  Interventions: Device: 50% AAB plus 50% autologous bone

INTERVENTIONS:
Device: 50% AAB plus 50% autologous bone — All patients were evaluated clinically and their medical histories were recorded. Preliminary screening, including the acquisition of intraoral and panoramic radiographs, was performed to evaluate potential patients' eligibility. Patients who met the selection criteria received oral hygiene instructions and debridement, if required, after which bone volumes were analysed using cone-beam computed tomography (CBCT; Imaging Sciences International, Hatfield, PA, USA).
  A staged approach was carried out at all sites. Thus, sinus lift grafting procedures were followed by implant placement 7-8 months later.
  Both groups received tapered implants with an anodised surface.
  Other Names: Bioss, Geistlisch Pharma AG, Wolhusen, Switzerland; Nobel Replace Tapered Groovy implant with Replace Select connection (Nobel Biocare®, Sweden)
  Arms: 50% AAB plus 50% autologous bone
Device: 100% AAB — All patients were evaluated clinically and their medical histories were recorded. Preliminary screening, including the acquisition of intraoral and panoramic radiographs, was performed to evaluate potential patients' eligibility. Patients who met the selection criteria received oral hygiene instructions and debridement, if required, after which bone volumes were analysed using cone-beam computed tomography (CBCT; Imaging Sciences International, Hatfield, PA, USA).
  A staged approach was carried out at all sites. Thus, sinus lift grafting procedures were followed by implant placement 7-8 months later. Both groups received tapered implants with an anodised surface.
  Other Names: Bioss, Geistlisch Pharma AG, Wolhusen, Switzerland; Nobel Replace Tapered Groovy implant with Replace Select connection (Nobel Biocare®, Sweden)
  Arms: 100% AAB

SUMMARY:
Background: Maxillary sinus floor augmentation is a standard surgical procedure to increase bone height in the atrophic posterior maxilla for dental implant placement. In bone reconstructive surgery, in general, autogenous bone is considered as the gold standard, primarily due to its osteogenic potential and remodelling capacity. Bone substitutes are available that can overcome the limitations of autologous bone due to their osteoconductive properties and biocompatibility. Several studies seem to validate these concepts, but further comparative trials are needed.

Aim: To compare the outcome of implants inserted in maxillary sinuses augmented with bovine bone grafts vs 50% bovine bone graft and 50% autologous bone according to a lateral approach.

Material and Methods: This study was designed as a randomised, controlled, clinical trial. Sixteen partially or fully edentulous patients, 20 sinuses, (four patients have been bilaterally treated) having 1 to 4 mm of residual crestal height below the maxillary sinuses were randomised according to a parallel group design. Sinuses were grafted according to a lateral approach. Group A (10 sinuses) was grafted with 50% anorganic bovine bone (Bio-Oss) and 50% autogenous bone, group B (10 sinuses) was grafted with 100% anorganic bovine bone (Bio-Oss). According with a two stages approach, after 7 months a total of 32 implants (Nobel Replace tapered groovy) were inserted with an insertion torque between 35 and 45 Ncm. At same surgical procedure a sample of bone was harvested for histomorphometric analysis . All implants were delayed loaded with screw retained temporary crowns 3 months after implants insertion and with screw retained definitive crowns 4 months later. Outcome measures were implant survival, biological and prosthetic complications, radiographic marginal bone-level changes, PPD and BOP. Clinical data were collected at baseline 6,12 months. Statistical significance was tested at the 0.05 probability level, and all values were presented as mean and standard deviation.

ELIGIBILITY:
Inclusion Criteria:

* Need for implant-supported prosthesis in maxillary posterior area.
* Need to insert implant in atrophic posterior maxilla, with a residual alveolar bone height 1 4 mm.
* ≥ 18 years of age.
* Provided written informed consent.
* Smokers of fewer than 10 cigarettes per day.
* Absence of sinus cyst or active sinusitis.

Exclusion Criteria:

* General contraindications to implant surgery.
* Occluding dentition in the area intended for implant installation
* Periodontitis.
* Bruxism.
* Immunosuppression.
* Previous history of irradiation of the head and neck area.
* Uncontrolled diabetes.
* Heavy smoker (>10 cigarettes/day).
* Poor oral hygiene.
* Current or past treatment with bisphosphonates.
* Substance abuse.
* Psychiatric disorder.
* Inability to complete follow-up ≥1 year.
* Lactation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-02; Primary Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
IMPLANT SURVIVAL | up to 12 months
  The removal of implants was dictated by instability, progressive marginal bone loss, infection, or implant fracture. The stability of individual implants was measured by the prosthodontist at the time of definitive crown delivery (5 months after implant placement) by applying 35 Ncm of removal torque. After 1 year, implant stability was tested manually with two dental mirror handles.

SECONDARY OUTCOMES:
MARGINAL BONE LEVELS | Baseline, 12 months
  Peri-implant marginal bone levels were evaluated on intraoral digital radiographs taken with the parallel technique. A blinded radiologist (FG), unaffiliated with the study centre, interpreted all radiographs. The distances from the mesial and distal interproximal bone to the reference point (the horizontal interface between the implant and abutment) were measured with a software tool (NIH Scion Image, ver. 4.0.2, Frederick, MD, USA) calibrated against the space between two threads to the nearest 0.1 mm, and the mean of these two measurements was calculated for each implant. The measurements were recorded with reference to the implant axis.

OTHER OUTCOMES:
MUCOSAL RESPONSE | Baseline, 12 months
  Probing pocket depth (PPD) and bleeding on probing (BOP) were measured by a blinded operator (AD) with a periodontal probe (PCP-UNC 15, Hu-Friedy Manufacturing) at 6 and 12 months. Three vestibular and three lingual values were collected for each implant by the same dentist.

CONTACTS AND LOCATIONS:
Overall Officials: Silvio M Meloni, DDS, Phd, MS, Principal Investigator — Università degli Studi di Sassari
Locations (1):
- Dipartimento di Scienze chirurgiche microchirurgiche e mediche dell'università degli studi di sassari, Sassari, SS, Italy